CLINICAL TRIAL: NCT06242158
Title: The 5-step Mini-open Method of Massive Rotator Cuff Repair and Clinical and Radiological Outcome
Brief Title: 5 Step Mini-open Method of Massive Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, PI, Kasr El Aini Hospital
Other Study IDs: MS-518-2019
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Massive Rotator Cuff Tears

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case with massive rotator cuff tear: Case with massive rotator cuff tear defined as more than 2 complete tendon tear that is repairable
  Interventions: Procedure: arthroscopic assisted mini-open 5 step repair

INTERVENTIONS:
Procedure: arthroscopic assisted mini-open 5 step repair — First step Identifying the tear size , quality and if reducible on the foot print . minimal removal of the bursa and pulling of the tendon with a grasper to reach the foot print area with gentle mobilization of the tendon .
  Step two Acromioplasty Using a probe, the LHBT was palpated and mobilized, looking for any signs of degeneration and fraying or instability . The LHBT was inspected either through the tear by the subacrominal portal or through the glenohumeral portal .
  Step three Antero-lateral mini-open approach was used through a longitudinal 4 cm skin incision Step four Transosseous repair using the giant needle was used. 3 to 4 number two fiber wire sutures was passed equidistance through the tendon Step five The subarominal bursa was used for biological augmentation of the repair

SUMMARY:
48 patients with massive rotator cuff tears were treated with a standardized five step technique of arthroscopic guided mini-open tranosseous repair with bursal augmentation. Their follow up is noted

DETAILED DESCRIPTION:
48 patients with massive rotator cuff tears were treated with a standardized five-step technique of arthroscopic guided mini-opentranosseous repair with bursal augmentation . ( 22 ) males and ( 26 ) females. age had a range of (58-68 ) with a mean (of 61 ) . The rt side was involved in ( 22 ) the lt side was involved in (26 ) . (12 ) patients had diabetes while one was on dialysis.

All patients were evaluated clinically for the range of movements of the shoulder in foreword flexion, abduction, ext, and int rotation. The constant score and UCLA scores were used for functional evaluation. Patients with flexion less than 90% were included in the study.

Standard plain x-ray of the shoulder and MRI were performed for all patients to evaluate the CSA and the condition of the rotator cuff. Tears were considered Massive rotator cuff tears if two or more tendons were involved. The degree of fatty degeneration and retraction of the tendon was not a contraindication for repair.

Surgical approach The procedures were performed under general anesthesia in association with interscalene brachial plexus block. The patient was positioned on a beach chair and conventional portals were used for both glen humeral and subacromial space.

First step Identifying the tear size, quality, and if reducible on the footprint. minimal removal of the bursa and pulling of the tendon with a grasper to reach the footprint area with gentle tendon mobilization. if the tendon is of bad quality and friable with the application of the grasper or if it is nonreducible on the footprint we stop the procedure of repair and shift to tendon transfer.

Step two Acromioplasty with removing the anterior and lateral part of the acromion in type 2,3 so we can reach a wide space allowing the blunt trocher 4mm diameter to slide comfortably in different positions of shoulder abduction. minimal removal of coracoacrominalligement was done to prevent superior instability .mimimal removal of the fibers of the deltoid anterior to prevent detachment of the anterior fibers of the deltoid when performing anterior lateral mini-open approach.

Using a probe, the LHBT was palpated and mobilized, looking for any signs of degeneration and fraying or instability. The LHBT was inspected either through the subacromial portal tear or the glenohumeral portal.

For patients aged 65 years or older, a tenotomy was performed. Tenodesis was performed on younger and active patients. Tenotomy was performed close to the origin of the glenoid labrum. Tenodesis, when indicated, was performed using fixing nonabsorbable sutures to the insertion pectoralis tendon by a separate incision.

Lastely the footprint is prepared at a slow speed bear with special consideration to localize and prepare the whole length and breadth of the footprint.

Step three Antero-lateral mini-open approach was used through a longitudinal 4 cm skin incision in line with anterior acromion and splitting the anterolateral raphe of the deltoid muscle between the anterior and middle fibers. A blunt deltoid retractor was applied and involvement and configuration of the torn tendon was confirmed by rotating the arm and attempting anatomical reduction on the footprint. A Cobb dissector was used to further mobilize the tendon passing deep under the acromion and pushing gently the rotator tendon to the outside towards the greater tuberosity bone Step four Transosseous repair using the giant needle was used. 3 to 4 number two fiber wire sutures were passed equidistance through the tendon (fig ). The giant needle was introduced to penetrate the bone at equidistance of the footprint and emerged from the skin about 5 cm from the tip of the greater tuberosity. A right angle hook was used superficially to the bursa to retrieve the distance end of the sutures. Before tightening the sutures the subacrominal bursa was mobilized gently from medial and posterior towards the tendon ends.

Step five The subacromial bursa was used for biological augmentation of the repair by overlapping the site of repair of the tendon to the bone. This was done by applying the sliding knot involving both the bursa and the tendon. Tighting the sutures pulls the tendon down on the bone and overlaps the bursa on the healing sight (fig ).

Post-operative The patient Weard an abduction brace and began pendulum and passive range-of-motion exercises one day after surgery. They began active range-of-motion exercises six weeks after surgery, muscle-strengthening exercises at three months, and occupational or sports activities at six months.

ELIGIBILITY:
Inclusion Criteria:

* a case with massive rotator cuff tear that is repairable (judged intraoperative by arthroscope that the tear returns to its footprint)
* ages from 60 to 84

Exclusion Criteria:

* Osteoarthritis
* associated fractures
* younger than 60 orolder than 84

Ages: 60 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: These are patients who presented to cairo university hospitals between 2019 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Constant score | (Pre operative) then at post operative 1 year and 2 years
  for function of shoulder

SECONDARY OUTCOMES:
Vas score | (Pre operative) then at post operative 1 year and 2 years
  for pain
UCLA score | (Pre operative) then at post operative 1 year and 2 years
  for function

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital - Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes